CLINICAL TRIAL: NCT02015065
Title: Phase II Trial of Vandetanib (ZD6474, Caprelsa(R) in Children and Adults With Wild-Type Gastrointestinal Stromal Tumors
Brief Title: Phase II Trial of Vandetanib in Children and Adults With Wild-Type Gastrointestinal Stromal Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brigitte Widemann, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130208; 13-C-0208
Record Dates: First submitted 2013-12-14; First posted 2013-12-19 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: GIST
Keywords: GIST; Small Molecule; Mesenchymal Tumor; Receptor Tyrosine Kinase; Survival
MeSH Terms: interventions — vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vandetanib in Children (Experimental): Children with measurable localized or metastatic wt-GIST
  Interventions: Drug: Vandetanib
- Vandetanib in Adults (Experimental): Adults with measurable localized or metastatic wt-GIST
  Interventions: Drug: Vandetanib

INTERVENTIONS:
Drug: Vandetanib — Vandetanib administered orally once per day continuously using a 28 day cycle until disease progression or unacceptable toxicity

SUMMARY:
Background:

-Some people with wild-type gastrointestinal stromal tumors (WT-GIST) have a deficiency in one of their proteins called succinate dehydrogenase (SDH). Vandetanib is a cancer drug that has been approved to treat thyroid cancer and has been used with some success in other tumors that have a similar loss of SDH. Researchers want to see if this drug can also decrease tumor growth in people with WT-GIST.

Objectives:

-To test whether the study drug will benefit people with WT-GIST.

Eligibility:

-Adults and children 3 years old and older with WT-GIST.

Design:

* Researchers will test participants tumor tissue to confirm it is the wild type of GIST.
* Participants will be screened with a medical history, physical exam, and blood tests. They will also have electrical recording of the heart (Eastern Cooperative Oncology Group (ECOG)) and scans of the tumor.
* Participants will take the study drug in 28-day cycles. Their doctor will decide how many cycles they can complete.

  * They will take the study drug once every day and record it in a diary.
  * On Day 14, they will also visit their doctor to look for side effects.
* Before cycles 2, 3 and 4, participants will have a physical exam, urine tests, blood pressure check, and blood tests. These tests will then be done periodically for as long as they are in the study.
* Before cycle 4, scans will be done to check the size of the cancer. Most of these will be repeated every 3-6 cycles.
* When they stop taking the study drug, participants will return to the clinic for a physical exam and blood tests.

DETAILED DESCRIPTION:
Background:

* Gastrointestinal stromal tumors (GISTs) are the most common mesenchymal tumor of the gastrointestinal tract, resistant to cytotoxic chemotherapy and radiation therapy. KIT and platelet derived growth factor receptor alpha (PDGFRA) mutations have been identified as tumor initiating events in 85% of adult patients with GIST, but 85% of GISTs in pediatric patients lack KIT and PDGFRA mutations (wild-type) and imatinib is not as effective in eliciting objective responses.
* Recent work in the Pediatric and Wild-Type (wt) GIST Clinic at the National Cancer Institute (NCI) led to the identification of succinate dehydrogenase (SDH) germline mutations in 12% patients with wt-GIST (6/34). SDH protein expression evaluated using immunohistochemistry (IHC) was markedly decreased or absent in 18/18 patients with pediatric wt-GIST. Thus the majority of wt-GIST are SDH-deficient. Vandetanib (ZACTIMA; ZD6474; AstraZeneca) is an oral small molecule antineoplastic drug that inhibits vascular endothelial growth factor receptor 2 (VEGFR2), estimated glomerular filtration rate (EGFR), and rearranged during transfection (RET)-dependent signaling. Preliminary preclinical data demonstrate marked growth inhibition of SDH-mutant/deficient renal cell carcinoma cell lines when treated with vandetanib.

Objective(s):

-Primary: To assess the clinical activity (radiographic response Response Evaluation Criteria in Solid Tumors (RECIST v1.1) of vandetanib in children and adults with wt-GIST using RECIST (v1.1).

Eligibility:

-Adults and children with measurable localized or metastatic wt-GIST confirmed in a Clinical Laboratory Improvement Amendments (CLIA) laboratory will be eligible for trial participation. Patients must have measurable disease by RECISTv1.1 and adequate organ function.

Design:

* This phase II trial will determine whether daily oral vandetanib is active in patients with wt-GIST. Vandetanib activity will be assessed primarily by radiographic response of measurable disease using RECISTv1.1.
* Vandetanib will be administered orally once daily continuously in the absence of toxicity or disease progression, using a 28-day cycle.
* Patients will be carefully monitored for toxicity and response. A small, optimal two-stage phase II design with a target response rate of 25% will be used. Nine evaluable patients will be enrolled initially. If 1 or more of the first 9 have a response, then accrual would continue until a total of 24 patients have enrolled. If there are 3 or more responses in 24 (12.5% or more) patients, then this would be sufficiently interesting activity to warrant further study.

ELIGIBILITY:
-INCLUSION CRITERIA

Age:

-greater than or equal to 3 years of age and Body Surface Area (BSA) greater than or equal to 0.5 m(2)

Diagnosis

* Histologically or cytologically confirmed Gastrointestinal Stromal Tumors (GIST) by the Laboratory of Pathology, National Cancer Institute (NCI).
* Absence of Kit and platelet derived growth factor receptor alpha (PDGFRA) mutation confirmed in a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory.
* Participants must have measurable disease as defined in Response Evaluation Criteria in Solid Tumors (RECIST (v1.1) as the presence of at least one lesion not previously irradiated, that can be accurately measured at baseline greater than or equal to 10mm in the longest diameter (except lymph nodes which must have short axis greater than or equal to 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.

Prior therapy:

There are no standard chemotherapy regimens known to be effective for wt-GIST. Therefore, previously untreated participants are eligible if their tumor(s) are measurable.

* Participants must be at least 4 weeks from prior surgical procedures and surgical incisions must be healed.
* Participants must have had their last fraction of external beam radiation therapy at least 4 weeks prior to enrollment.
* Participants must have had their last dose of cytotoxic chemotherapy at least 28 days prior to enrollment, their last dose of biological therapy, such as biological response modifiers (e.g., cytokines), immunomodulatory agents, vaccines, differentiating agents, used to treat their cancer at least 7 days prior to enrollment, their last dose of a monoclonal antibody at least 30 days prior to enrollment, and their last dose of any investigational agent at least 30 days prior to enrollment.
* Participants must have received their last dose of short acting colony stimulating factor, such as filgrastim or sargramostim at least 72 hours prior to enrollment and their last dose of long-acting colony stimulating factors, such as PEG-filgrastim at least 7 days prior to enrollment.
* Participants must have recovered from the acute toxic effects of prior therapy to a grade 1 (Common Terminology Criteria in Adverse Events (CTCAE v.4.0)) level prior to enrollment (does not apply to alopecia).

Performance Status: Lansky (for participants 10 years of age or younger) or Karnofsky (for participants older than 10 years) performance score greater than 50

Patients must have normal organ and marrow function as defined below:

* Hematological Function: The peripheral absolute neutrophil count must be at least 1,500/microL and the platelet count must be at least 100,000/microL within 72 hours prior to enrollment.
* Coagulation: Prothrombin Time (PT) and Partial Thromboplastin Time (PTT) must not be more than 1.5 x upper limit of normal (ULN) within 72 hours prior to enrollment. PT and PTT should drawn by venipuncture, rather than from a central venous catheter when feasible.
* Hepatic Function: Bilirubin must not be more than 1.5 x ULN (does not apply to patients with Gilberts Disease) and the aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must not be more than 2.5 x ULN within 72 hours prior to enrollment, or greater than 5.0 X ULN if in the Investigator s judgment it is related to liver metastases. AST and ALT may be up to 5 x ULN within 72 hours prior to enrollment in participants with hepatic metastases.
* Renal Function: Participants must have an age-adjusted normal serum creatinine (see Table) or a creatinine clearance of at least 50 ml/min/1.73 m(2).

Age (years) Male Female

3 to 5 = .42

5 to <10 = 1

10 to <13 = 1.2

13 to <16 = 1.5 male and 1.4 female

16 and older = 1.7 male and 1.4 female

Hypertension:

-Participants should have normal blood pressure according to age. Participants 18 years of age and younger should have a blood pressure 95th percentile for age, height and gender, and should not be receiving medication for treatment of hypertension. Preexisting hypertension in adults should be controlled (either with pharmacological or non-pharmacological methods) at the time of enrollment.

Birth Control:

* Participants of child-bearing or child-fathering potential must be willing to use a medically effective form of birth control, which includes abstinence, while taking vandetanib and for 4 months after the last dose. [Female patients must be 1 year postmenopausal, surgically sterile, or using an acceptable method of contraception (an acceptable method of contraception is defined as a barrier method in conjunction with a spermicide) for the duration of the study (from the time they sign the informed consent form [ICF]) and for 3 months after the last dose of vandetanib to prevent pregnancy. In addition, oral contraceptives, approved contraceptive implant, long-term injectable contraception, intrauterine device, or tubal ligation are allowed. Oral contraception alone is not acceptable; additional barrier methods in conjunction with spermicide must be used.
* Male patients must be surgically sterile or using an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) for the duration of the study (from the time they sign the ICF) and for 4 months after the last dose of vandetanib to prevent pregnancy in a partner.]
* Negative pregnancy test for women of childbearing potential.

Informed Consent:

-Participants who are greater than or equal to 18 years of age or Legally Authorized Representative (LAR) of participants who are younger than 18 years must sign an informed consent for the Pediatric Oncology Branch (POB) Screening Protocol (01-C-0157: Eligibility Screening and Tissue Procurement for the National Cancer Institute (NCI), Pediatric Oncology Branch (POB) Clinical Research Protocols) prior to participating in studies required to determine eligibility for this trial. After confirmation of eligibility, participants who are greater than or equal to 18 years of age or LAR of minor participants must sign an informed consent document for this trial, indicating that they are aware of the investigational nature of the proposed treatment, the risks and benefits of participating and the alternatives to participating, prior to the conduct of any study procedures.

EXCLUSION CRITERIA

Presence of any of the following will prevent a subject from participation:

* Pregnant or breast feeding females because vandetanib may be harmful to the developing fetus or nursing infant and has been found to be embryotoxic, fetotoxic and teratogenic in rats.
* Subjects who are receiving any other investigational agents or who have received an investigational agent within 28 days prior to enrollment (does not apply to participation in survival follow up), or who have previous exposure to vandetanib.
* Abnormal Electrolyte Levels: Participants with a serum potassium less than 3.5 mmol/L or a serum ionized calcium or magnesium below the lower limits of normal (or above Common Terminology Criteria in Adverse Events (CTCAE) Grade 1 upper limit). Correction of these electrolyte abnormalities with supplements is allowed. (Serum calcium above the CTCAE Grade 1 upper limit. In cases where the serum calcium is below the normal range, the calcium adjusted for albumin is to be obtained and substituted for the measured serum value. Exclusion is to then be based on the calcium adjusted for albumin values falling below the normal limit: Corrected Calcium = Ca + 0.8 x (4-serum albumin).)
* Presence of hypertension: Diastolic blood pressure above the 95% for age in children (Appendix 2) and > 160 mmHg systolic or >100 mmHg diastolic in adults on at least 2 of 3 measurements with an appropriate-size cuff who are unable to achieve blood pressure control with optimal anti-hypertensive therapy. Patients who are treated with antihypertensive medications with good response are eligible.

History of Cardiac Disorder:

* Participants with a history of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia, uncontrolled atrial fibrillation, left bundle branch block) that is symptomatic or requires treatment (except for controlled atrial fibrillation).
* History of any significant cardiac event (e.g. myocardial infarction), superior vena cava syndrome, New York Heart Association (NYHA) classification of heart disease greater than or equal 2 within 12 weeks before starting treatment, or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
* Participants with a history of congenitally prolonged corrected QT interval (QTc), a first degree relative with unexplained sudden death under 40 years of age, or a measured QTcB (Bazetts correction) longer than 480 msec on electrocardiography (ECG). ECGs should be performed after correction of electrolyte abnormalities. Participants with a prolonged QTcB should have a repeat ECG twice, at least 24 hour apart, and the average of the 3 QTcBs should not exceed 480 msec. History of QT prolongation associated with other medications that required discontinuation of that medication.
* Participants receiving a medication that has a known risk of QTc prolongation or is associated with Torsades de Pointes or any prohibited medications, concomitantly or within 14 days (28 days for levomethadyl) of enrollment.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of vandetanib as evidenced by uncontrolled nausea, vomiting or diarrhea and/or current need for parenteral support with iron or Vitamin B.
* Other clinically severe or uncontrolled systemic illness or any concurrent condition that in the view of the principal investigator could compromise the participant's ability to tolerate vandetanib or could compromise study procedures or endpoints, including interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease.
* Unstable brain metastases or spinal cord compression that requires treatment, unless the treatment ended at least 4 weeks before starting treatment and the condition has been stable without steroid treatment for at least 10 days.
* Major surgery (includes surgery that carries significant risk of blood loss, extended periods of general anesthesia, or requires at least an overnight hospital admission) within 28 days before starting treatment.
* Involvement in the planning and/or conduct of the study.
* Previous enrollment in the present study.
* Previous or current malignancies of other histologies within the last 5 years, with the exception of in situ carcinoma of the cervix and adequately treated basal cell or squamous cell carcinoma of the skin.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-12-14 (Actual); Primary Completion 2016-05-04 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0208.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to lack of efficacy no participants were enrolled in Dose Level 150mg/m^2 Vandetanib Pediatric Arm/Group.
Groups:
- 200 mg Vandetanib Adult: Initially patients 18 years and older at the time of enrollment on this study will start vandetanib at a fixed dose of 200 mg once daily (QD) for cycles 1, 2, and 3. One cycle = 28 days. If vandetanib was tolerated at 200mg daily the dose was increased to 300mg daily. Because of excessive toxicity at the 300mg daily dose the study was amended to maintain a dose of 200mg daily in patients 18 years and older after cycle 3.
- 300 mg Vandetanib Adult: Patients 18 years and older at the time of enrollment on this study will start vandetanib at a fixed dose of 200 mg once daily (QD) for cycles 1, 2, and 3. One cycle = 28 days.
  If Vandetanib was well tolerated: Cycles ≥4: 300 mg/dose
- Dose Level 100mg/m^2 Vandetanib Pediatric: Patients younger than 18 years of age at the time of enrollment were started at a dose of 100 mg/m^2 based on a dosing nomogram with a planned increase in the dose to 150mg/m^2/day after the third cycle if the drug was tolerated. One cycle = 28 days.
Period: Overall Study
Arm/Group | 200 mg Vandetanib Adult | 300 mg Vandetanib Adult | Dose Level 100mg/m^2 Vandetanib Pediatric
Started | 2 | 5 | 2
Completed | 1 | 3 | 1
Not Completed | 1 | 2 | 1
Not completed — Death on study | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 200 mg Vandetanib Adult | 300 mg Vandetanib Adult | Dose Level 100mg/m^2 Vandetanib Pediatric | Total
Number analyzed (Participants) | 2 | 5 | 2 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 2 | 2
  Between 18 and 65 years | 2 | 5 | 0 | 7
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (3.0) | 34.3 (13.17) | 13.2 (2.12) | 27.42 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 2 | 7
  Male | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not meeting definition for Hispanic or Latino | 2 | 5 | 1 | 8
  Mexican, Puerto Rican, Cuban, Central or So. Amer. | 0 | 0 | 1 | 1
  Black or African American | 1 | 0 | 0 | 1
  White | 1 | 5 | 0 | 6
  Asian | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 5 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinical Activity-radiographic Response
Description: Clinical activity will be assessed primarily by radiographic response of measurable disease using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete Response is disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study); (Note: the appearance of one or more new lesions is also considered progressions). Stable Disease is neither sufficient shrinkage to qualify for Partial Response nor sufficient increase to qualify for Progressive Disease, taking as reference the smallest sum diameters while on study.
Time Frame: Every 3 cycles x4 and then every 6 cycles (1 cycle = 28 days) until removal from protocol therapy, an average of 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | 200 mg Vandetanib Adult | 300 mg Vandetanib Adult | Dose Level 100mg/m^2 Vandetanib Pediatric
Number analyzed (Participants) | 2 | 5 | 2
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0
  Stable Disease | 1 | 2 | 1
  Progressive Disease | 1 | 3 | 1

2. Secondary Outcome: Count of Participants With Serious and Non-serious Adverse Events
Description: The count of participants with serious and non-serious adverse events was assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 32 months and 1 day.
Measure: Count of Participants; unit: Participants
Arm/Group | 200 mg Vandetanib Adult | 300 mg Vandetanib Adult | Dose Level 100mg/m^2 Vandetanib Pediatric
Number analyzed (Participants) | 2 | 5 | 2
Participants | 2 | 5 | 2

3. Secondary Outcome: Percentage of Participants Overall Survival
Description: Overall survival is defined as the date of on-study to the date of death from any cause or last follow up.
Time Frame: Overall survival was computed using the number of months from the date of on study to the date of death, an average of 12 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 200 mg Vandetanib Adult | 300 mg Vandetanib Adult | Dose Level 100mg/m^2 Vandetanib Pediatric
Number analyzed (Participants) | 2 | 5 | 2
percentage of participants | 50 [0.6 to 91] | 60 [12.6 to 88.2] | 50 [0.6 to 91]

4. Secondary Outcome: Progression Free-Survival
Description: Progression free survival is defined as the time interval from start of treatment to documented evidence of disease progression. Disease progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: Patients will be evaluated approximately 60 days after last dose of investigational drug until removal of protocol therapy, an average of 12 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 200 mg Vandetanib Adult | 300 mg Vandetanib Adult | Dose Level 100mg/m^2 Vandetanib Pediatric
Number analyzed (Participants) | 1 | 5 | 2
Months | 4 [0.6 to 91] | 5.1 [1.8 to 22.5] | 13.4 [2.7 to 24.1]

5. Secondary Outcome: Maximum Standardized Uptake Value (SUVmax) on Fluorodeoxyglucose Positron Emission Tomography (FDG-PET)
Description: The maximum standardized uptake value (SUVmax) was used to measure the uptake of FDG-PET by the Gastrointestinal Tumors.
Time Frame: Baseline and at a subsequent PET performed on or about day 3-6 of cycle 1
Population: Data were only collected from patients >/= 15 years of age.
Measure: Median (Full Range); unit: g/mL
Arm/Group | 200 mg Vandetanib Adult | 300 mg Vandetanib Adult | Dose Level 100mg/m^2 Vandetanib Pediatric
Number analyzed (Participants) | 1 | 3 | 0
g/mL
  Baseline | 22.4 [22.4 to 22.4] | 21.4 [15.6 to 30.7] |
  Day 3-6 of cycle 1 | 22.0 [22.0 to 22.0] | 12.4 [7.5 to 19.3] |

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 32 months and 1 day.
Arm/Group | 200 mg Vandetanib Adult | 300 mg Vandetanib Adult | Dose Level 100mg/m^2 Vandetanib Pediatric
All-Cause Mortality (participants affected / at risk) | 1/2 | 2/5 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 4/5 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 5/5 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg Vandetanib Adult (N=2) | 300 mg Vandetanib Adult (N=5) | Dose Level 100mg/m^2 Vandetanib Pediatric (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg Vandetanib Adult (N=2) | 300 mg Vandetanib Adult (N=5) | Dose Level 100mg/m^2 Vandetanib Pediatric (N=2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 4 (6) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 2 (4) | 4 (6) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 2 (3)
Weight loss (Investigations) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (21) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (2) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 4 (9) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, not clinically significant (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (6) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Heaviness in the legs.
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (10) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Psychiatric disorders) | 0 (0) | 4 (7) | 0 (0)
Psychiatric disorders - Other, hypomanic (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 3 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Skin and subcutaneous tissue disorders - itchiness/redness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT02015065/Prot_SAP_000.pdf
  • Informed Consent Form: Standard consent (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT02015065/ICF_001.pdf
  • Informed Consent Form: Parent QOL consent (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT02015065/ICF_002.pdf